CLINICAL TRIAL: NCT00136253
Title: Overcoming Nutritional Barriers in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: DK51472
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2005-12-13 (Estimated); Status verified 2004-10

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

INTERVENTIONS:
Behavioral: Help dietitians and patients address specific nutritional barriers

SUMMARY:
American hemodialysis patients are frequently malnourished. This contributes to dialysis patient mortality rates that are the highest in the industrialized world at 22% per year. Poor nutritional status probably also contributes to high health care costs (an average of two hospitalizations annually per patient and total Medicare expenditures of $11 billion per year) and diminished quality of life. The researchers' prior work identified several potentially modifiable nutritional barriers (e.g. poor appetite, inadequate dialysis dose, poor nutritional knowledge, low fluid intake, and needing help shopping and cooking) and pilot tested a promising approach to overcome these barriers.

This proposed community-based randomized controlled trial extends the researchers' prior work by targeting specific nutritional barriers with a tailored feedback and education intervention. Approximately 40 dialysis facilities in northeast Ohio will be randomly assigned to intervention and control groups, with approximately 100 malnourished patients enrolled from 20 intervention facilities and 100 from 20 control facilities. Baseline evaluation will include measures of nutritional status, specific barriers, inpatient expenditures, and quality of life. On a monthly basis for 12 months, intervention patients and their dietitians will receive tailored feedback and education on overcoming patient-specific barriers. They will then meet monthly to jointly formulate a care plan addressing these barriers. Control patients will continue to get usual care. Major analyses will compare changes in nutritional parameters in intervention vs. control patients with adjustment for nesting of patients within facilities.

The proposed project will test a novel intervention that targets patients and providers as they together make nutrition-related decisions. Overcoming specific barriers may lead not only to improved nutritional status but also to better patient survival, decreased health care costs, and increased quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Most recent albumin and mean albumin over last 3 months <3.7 g/dL by bromcresol green method (or <3.4 g/dL by bromcresol purple method)
* Age greater than or equal to 18 years
* On chronic hemodialysis at least 9 months

Exclusion Criteria:

* Mentally incompetent
* Cirrhosis
* AIDS
* Cancer
* Terminal illness
* Malabsorption
* Receiving total parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-02; Study Completion 2004-10

PRIMARY OUTCOMES:
Change in albumin
Change in albumin of 0.20 or greater and survival

SECONDARY OUTCOMES:
Change in subjective global assessment, weight, dietary intake, specific nutritional barriers

CONTACTS AND LOCATIONS:
Overall Officials: Ashwini Sehgal, MD, Principal Investigator — MetroHealth Medical Center